CLINICAL TRIAL: NCT04351594
Title: Effect of a Menthol Gel (Biofreeze) on the Symptoms Associated with Knee Osteoarthritis: a Double-blind Randomized Control Trial.
Brief Title: Biofreeze and the Effect on Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Nick Smith, Dr. Nicholas Smith MD, MSc, FRCSC, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MUN8051
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Pain management; Menthol; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Agnosia | interventions — Gels; Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical analgesia (+Menthol) (Experimental): Biofreeze Topical Gel with active ingredient (Menthol 4%)
  Interventions: Drug: Biofreeze 4 % Topical Gel
- Topical analgesia (-Menthol) (Placebo Comparator): Biofreeze Topical Gel with no active ingredient (Menthol 0%)
  Interventions: Other: Biofreeze placebo gel

INTERVENTIONS:
Drug: Biofreeze 4 % Topical Gel — Biofreeze gel with active manufactured ingredient (Menthol 4%)
  Other Names: Menthol 4% Topical gel
  Arms: Topical analgesia (+Menthol)
Other: Biofreeze placebo gel — Biofreeze gel with no active manufactured to have the same look, feel and odour as Biofreeze topical gel.
  Other Names: Placebo gel (Menthol 0%)
  Arms: Topical analgesia (-Menthol)

SUMMARY:
Knee osteoarthritis (OA) is a progressive disease that can be accompanied by considerable joint pain and dysfunction. It is a goal in the medical field to find effective treatments for knee OA that are non-interventional, have minor or no negative side effects, and are relatively easy to administer for the patient and health care professionals. Biofreeze, a topical analgesic containing menthol, is an easily accessible gel, with no known serious negative side effects. If the application of Biofreeze can reduce the pain and dysfunction associated with knee OA, it could be an effective treatment for patients. The objective of the study is to assess how 4 weeks of Biofreeze application to a knee affected by OA effects pain and dysfunction associated with the disease.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a disease which results in deterioration with articular cartilage and bone tissue of the knee joint (Felson et al., 2000). The disease is prevalent in the elderly and as it progresses, can cause serious joint pain and a lot of knee dysfunction (National Collaborating Centre for Chronic Conditions, 2008). In addition to surgical intervention, there are currently a multitude of non-surgical interventional treatments which have been used to help patients deal with the pain and dysfunction associated with OA. This includes exercise, weight loss, orthotics, topical and oral medications, therapeutic modalities and even more (Dadabo, Fram, and Jayabalan, 2019). While the aforementioned treatments all have advantages, there are some disadvantages including but not limited to; negative side effects of oral medications, exercise intolerance secondary to pain as well as risk of injury, difficulty in maintaining a healthy diet, cost associated with receiving therapeutic modalities, all of which could make the treatments impractical for some or all patients. It is a goal for health researchers, to discover a treatment which can significantly reduce pain and dysfunction associated with knee OA while also limiting the negative side effects or difficulties associated with using the treatment. There are a few studies which have looked at the effect of topical treatments on symptoms associated with knee OA. One study performed a double-blind, randomized, placebo-controlled clinical trial using linseed oil (Mosavat et al., 2018). This study found that the administration of linseed oil significantly reduced pain and other symptoms associated with knee OA compared to the control. Another study used a topical non-steroidal anti-inflammatory drug (NSAID) to treat knee OA pain (Bookman, Williams, and Shainhouse, 2004).This study also found that the treatment helped with pain, the drug was accompanied with some local skin irritation and minimal systemic side effects (Bookman et al.,2004). Biofreeze, a topical analgesic containing menthol, is a relatively cost-efficient item with no known adverse side effects. If the administration of Biofreeze to a knee affected with OA relieves pain and symptoms associated with OA, it could be a safe and effective treatment for knee OA patients to use. The primary objective in this study is to assess the affects of a menthol based topical agent on osteoarthritis of the knee. Outcome measures are based on scores obtained from the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC questionnaire is a patient-administered questionnaire that contains 24 questions, targeting areas of pain, stiffness and physical function, and can be completed in less than 5 minutes. The questionnaire will be given to the patients at the beginning and at the end of the 4 week study to compare differences.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 50-80 years
2. Body mass index (BMI) less than 40
3. Knee osteoarthritis of grade one or more according to Kellgren-Lawrence scale
4. Average pain intensity of grade 4 or more on a 10-point visual analogue scale for at least 6 months.
5. Meet clinical and radiographic criteria of the American College of Rheumatology (ACR) for knee OA

Exclusion Criteria:

1. Acute arthritis,
2. Rheumatologic diseases
3. Infective arthritis
4. Traumatic arthritis,
5. History of knee replacement surgery
6. Patients receiving multiple corticosteroid injections (Greater than 2 injections)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Efficacy comparison of (Biofreeze) Menthol 4%, Menthol 0% as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), version 3.0 | 4 weeks
  Endpoint is a non-inferiority statistical comparison. Comparison is based off of analysis of identical questionnaires administered at baseline and at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nick Smith, MD (FRCSC), Principal Investigator — Memorial University Orthopaedic Surgery
Locations (1):
- Memorial University, Faculty of Medicine Department of Surgery, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No
Investigators plan to share the study results as a whole but no plans to share individual results.

REFERENCES:
- [Background] Airaksinen OV, Kyrklund N, Latvala K, Kouri JP, Gronblad M, Kolari P. Efficacy of cold gel for soft tissue injuries: a prospective randomized double-blinded trial. Am J Sports Med. 2003 Sep-Oct;31(5):680-4. doi: 10.1177/03635465030310050801. PMID 12975186
- [Background] Bookman AA, Williams KS, Shainhouse JZ. Effect of a topical diclofenac solution for relieving symptoms of primary osteoarthritis of the knee: a randomized controlled trial. CMAJ. 2004 Aug 17;171(4):333-8. doi: 10.1503/cmaj.1031793. PMID 15313991
- [Background] Mosavat SH, Masoudi N, Hajimehdipoor H, Emami Meybodi MK, Niktabe Z, Tabarrai M, Ghorat F, Khodadoost M. Efficacy of topical Linum usitatissimum L. (flaxseed) oil in knee osteoarthritis: A double-blind, randomized, placebo-controlled clinical trial. Complement Ther Clin Pract. 2018 May;31:302-307. doi: 10.1016/j.ctcp.2018.03.003. Epub 2018 Mar 14. No abstract available. PMID 29705472
- [Background] Topp R, Brosky JA Jr, Pieschel D. The effect of either topical menthol or a placebo on functioning and knee pain among patients with knee OA. J Geriatr Phys Ther. 2013 Apr-Jun;36(2):92-9. doi: 10.1519/JPT.0b013e318268dde1. PMID 22976810